CLINICAL TRIAL: NCT02925559
Title: Effect of Anti-diabetic Drugs on Glycemic Variability. A Comparison Between Gliclazide MR (Modified Release) and Dapagliflozin on Glycemic Variability Measured by Continuous Glucose Monitoring (CGM) in Patients With Uncontrolled Type 2 Diabetes
Brief Title: Effect of Anti-diabetic Drugs on Glycemic Variability
Acronym: EFFORT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro de Diabetes Curitiba Ltda (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-14-10377
Record Dates: First submitted 2016-09-28; First posted 2016-10-06 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Glycemic Variability; Dapagliflozin; Gliclazide MR; Continuous Glucose Monitoring; Mean Amplitude of Glycemic Excursions; MAGE
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Gliclazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapagliflozin (Experimental): The active treatment will include a 10 mg dose of dapagliflozin orally once a day.
  Interventions: Drug: Dapagliflozin
- Gliclazide MR (Active Comparator): As comparator, gliclazide MR will be administered at a dose of 120 mg orally once a day.
  Interventions: Drug: Gliclazide MR

INTERVENTIONS:
Drug: Dapagliflozin — The active treatment will include a 10 mg dose of dapagliflozin orally once a day.
  Other Names: Farxiga; Forxiga
  Arms: Dapagliflozin
Drug: Gliclazide MR — As comparator, gliclazide MR will be administered at a dose of 120 mg orally once a day.
  Other Names: Diamicron MR
  Arms: Gliclazide MR

SUMMARY:
Objectives

Primary objective:

To access the change from baseline to week 12 in MAGE index of glycemic variability measured by CGMS for dapagliflozin versus. gliclazide MR.

Secondary objectives:

1. Change from baseline to week 12 in glycated hemoglobin A1c (HbA1c), fasting plasma glucose, postprandial glucose and achievement of HbA1c ≤6.5% and <7% at the end of the study) for dapagliflozin versus gliclazide MR.
2. Change from baseline to week 12 in glycemic variability defined by the interquartile range (IQR - interval between 25th and 75th percentiles) measured by CGMS for dapagliflozin versus gliclazide MR.
3. Change from baseline to week 12 in glycemic variability measured by the Standard Deviation of the mean glycemia (SD) measured by CGMS for dapagliflozin versus gliclazide MR.
4. Change from baseline to week 12 in glycemic variability measured by the Coefficient of Variation (CV) measured by CGMS for dapagliflozin versus gliclazide MR.
5. Change from baseline to week 12 in the time spent on hypoglycemic range (glycemia <70mg/dL) measured by CGMS for dapagliflozin versus gliclazide MR.

Study design This is a single-center, prospective, randomized, open-label, comparative, phase IV study to compare the effects of gliclazide MR and dapagliflozin on Glycemic Variability in patients with Type 2 Diabetes Mellitus (T2DM). All patients should be treatment naïve or receive standard of care therapy for T2DM as well as for co-morbidities based on accepted guidelines and local best practices.

Target patient population Approximately 120 patients with T2DM will be randomized from study site. Patients who were treated with metformin only and had inadequate glycemic control at the time of enrollment as well as treatment naïve or non-medically treated (e.g., diet) patients, will be enrolled and receive either dapagliflozin 10mg qd or comparator gliclazide MR 120mg qd in addition to standard of care treatment for T2DM and co-morbidities.

Investigational product, dosage and mode of administration Dapagliflozin 10mg tablets administered orally once daily for 12 weeks.

Comparator, dosage and mode of administration Gliclazide MR 60mg tablets administered orally, 2 tablets once daily for 12 weeks.

Duration of treatment The treatment with study medication or comparator will have a total duration of 15 weeks.

DETAILED DESCRIPTION:
INTRODUCTION Dapagliflozin is a highly potent, selective, and reversible inhibitor of sodium-glucose cotransporter-2 (SGLT2), the major transporter responsible for renal glucose reabsorption.1 Dapagliflozin lowers plasma glucose by inhibiting the renal reabsorption of glucose and by promoting its urinary excretion in patients with type 2 diabetes mellitus (T2DM).

Gliclazide MR is a highly potent and selective sulphonylurea considered by specialists a reference in this class, because of its low risk of hypoglycemia and no increasing in cardiovascular mortality. Gliclazide MR increases the physiological mechanism of insulin secretion, thus reducing the postprandial and fasting glucose levels in patients with type 2 diabetes.

There is an increasing large amount of evidences showing that rapid fluctuations in blood glucose and high glycemic variability may have an important role in the development of diabetes complications. Cardiovascular disease, endothelial dysfunction and oxidative stress are common complications among patients with type 2 diabetes and glycemic variability may be an important factor in their development. Previous studies have shown that vildagliptin, a dipeptidyl peptidase 4 inhibitor (DPP-4 inhibitor), could improve not only the mean blood glucose but also the 24-hour glucose fluctuation by restoring the physiological pattern of insulin and glucagon secretion. SGLT-2 inhibitors are novel anti-diabetic drugs and currently there are not published studies that evaluated their effects on glycemic variability calculated by the widely used methods like mean amplitude of glycemic excursion (MAGE), standard deviation of the mean glycemia (SD), coefficient of variation (CV) and interquartile range (IQR).

The aim of the current study is to compare the effect of gliclazide MR with dapagliflozin on the glycemic variability using a continuous glucose monitoring system (CGMS) to determine MAGE, SD, CV and IQR.

2. METHODOLOGY 2.1 Study Population (Target population of Clinical Trial Subjects) A total of 120 patients with documented Type 2 Diabetes will be enrolled, considering an expected screening failure rate of 30% (n=22) and an expected dropout rate of 8% (n=10), based in previous studies conducted in our center using similar populations and period. We estimate that 88 (44 in each group) subjects will complete all protocol procedures. Per-protocol analysis will be restricted to the participants who fulfill the protocol in terms of the eligibility, interventions and outcome assessment. To be as close to a real life scenario as possible, this clinical trial will include subjects patients who were treated with metformin only and had inadequate glycemic control at the time of enrollment as well as treatment naïve or non-medically treated (e.g., diet) patients.

2.2 Investigational Product, Posology and Method of Administration The active treatment will include a 10 mg dose of dapagliflozin orally once a day.

2.3 Comparator, Posology and Method of Administration As comparator, gliclazide MR will be administered at a dose of 120 mg orally once a day.

2.4 Study Duration The study will have an expected total duration of 15 months (12 months for recruitment and 12 weeks of active treatment).

2.5 Methods and Assessments Patients will be randomized after revision of inclusion and exclusion criteria. Randomization will occur in a 1:1 manner using a validated computerized system until completion of 88 randomized patients.

Patients from group 1 (n~44) will receive the study medication (dapagliflozin) and the ones from Group 2 (n~44) will receive the comparator gliclazide MR on top of usual treatment for type 2 diabetes. Treatments with the study medication or comparator will last 12+/-1 weeks. All patients for both groups will receive the same guidelines about the diet (caloric and macronutrient contents) and physical activity by the same dietitian from the study site at the beginning of study. A "blinded to the patient" Continuous Glucose Monitoring System (CGMS, iPro2 (TM) with Enlite-Sensor (TM); Medtronic Mini-Med Inc., Northridge, California, USA) will be inserted subcutaneously. The sensor is a glucose oxidase-based platinum electrode that is inserted through a needle into the subcutaneous tissue of the anterior abdominal wall and allows up to 288 glucose readings per day. The CGMS will be placed for 72 hours at beginning (in the last three days of run-in phase) before starting the study medications and again at the end of the study in the last three days of the study treatment. The validated softwares Glyculator (TM) or EasyGV (TM) will calculate the glycemic variability parameters MAGE, SD and CV IQR will be calculated by the software Captür-AGP (TM). Biochemical markers of glycemic control (HbA1c, fasting glucose and postprandial glucose) will be determined at beginning and at the end of the treatment period. Each patient will maintain regular visits to his assistant doctor. At the end, the two groups will be compared according to the following parameters calculated based on results obtained on both CGMS tests, blood samples and patient Clinical Research Form (CRF)

* Glycemic variability parameters: MAGE, SD, CV and IQR
* Glycemic controls parameters: HbA1c, fasting glucose and postprandial glucose
* Exploratory variables: incidence of urinary tract Infection and genital infection and incidence of volume depletion.

2.6 Sample size and Statistical methods To determine the sample size and obtain a clinical and statistical significant result in the primary variable (difference >14.5mg/dL on glycemic variability), it was used MAGE (mean amplitude of glycemic excursion). As MAGE is glycemic amplitude measured in mg/dL, it was arbitrarily set a difference of ≥ 14.5, which may be clinically important for the patient as judged by the study center team and its expert consultants. There is not a good study of T2DM patients that establishes which MAGE difference or improvement could be significant to prevent diabetes complications.

Sample size was calculated based on the provided parameter: significance level (adjusted for sidedness) = 0.025, standard deviation for MAGE = 24mg/dL, power = 0.8, and a between-group difference in mean MAGE equal to 14.5 mg/dL. The variable calculated was the total number of patients. A total of 44 patients in each group (dapagliflozin 10 mg or gliclazide MR 120 mg) must complete this two-treatment parallel-design study. Considering an expected screening failure rate of 30% (n=11 per group) and an expected dropout rate of 8% (n=5 per group), based in previous studies in our center using similar populations and period, a total of 60 patients per group (120 total) will be enrolled.

Demographic and baseline characteristics will be represented by distributions of frequency and summarized statistics based on the dataset, both for each treatment group and all clinical trial subjects combined. The main baseline characteristics will be presented. ANCOVA will be used with adjustment for baseline values. For primary and secondary variables, all quantitative, it will be used Student's t-test or Mann-Whitney test for the statistical evaluation and comparison between groups. In all tests, it will be used the significance level of 5% or p<0.05.

2.7 Study Design and Rationale

This is a single-center, Prospective, Randomized, Open-label, Comparative, Phase IV Study to compare the effects of gliclazide MR and dapagliflozin on Glycemic Variability in patients with Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

A. Informed consent form obtained before any study-related activity. Study-related activities are any procedure that would not be performed during the normal treatment of the patient.

B. All study subjects must be patients diagnosed with type 2 diabetes based on current guidelines of Brazilian Society of Diabetes and/or American Diabetes Association (ADA) and they should have all the following criteria:

* Age ≥40 years old.
* HbA1c ≥7% at randomization.
* Drug naïve or metformin treated with a stable dose for at least 3 months.

Exclusion Criteria:

1. Acute vascular event (cardiac, cerebral or peripheral) for at least 2 months of randomization.
2. Patient on chronic dialysis and/or renal transplantation and/or serum creatinine >1.5 mg/dL and/or estimated glomerular filtration rate (eGFR) < 45ml/min (MDRD) and/or Creatinine Clearance <60ml/min.
3. Patients with HIV, severe autoimmune disease or chronic treatment with oral steroids (>30 consecutive days).
4. Current or previous treatment with any SGLT-2 inhibitor within 2 months prior to randomization.
5. Current or previous treatment with any type of insulin within 2 months prior to randomization.
6. Current or previous treatment with any sulphonylurea and meglitinide within 2 months prior to randomization.
7. Current or previous treatment with any DPP-4 inhibitor or glucagon-like peptide-1 (GLP-1) receptor agonist within 2 months prior to randomization.
8. Current or previous treatment with acarbose within 2 months prior to randomization.
9. Sustained arterial hypertension ≥160/100mm Hg.
10. Body mass index (BMI) >50 kg/m².
11. HbA1c ≥10.5% at randomization.
12. Transaminases (aspartate aminotransferase and/or alanine aminotransferase) >2.5 x upper limit of normal.
13. Total bilirubin >2.5 x upper limit of normal
14. Chronic liver disease or alcoholic liver disease.
15. LDL-cholesterol >250 mg/dL (>6.48 mmol/L).
16. Triglycerides >1000 mg/dL (>11.3 mmol/L).
17. HDL-cholesterol <25 mg/dL (<0.64 mmol/L).
18. Positive haematuria observed in urine sample obtained in the run-in visit.
19. Prescription of any investigational medication within 3 months before the screening visit.
20. Prescription of any investigational medication within the period between 3 months and one year before the screening visit (visit 1), unless there is a direct benefit to the study subject, at the discretion of the investigator.
21. Pregnant or breastfeeding patients.
22. Previous participation on this study.
23. Individuals at risk for poor adherence to the protocol or medication.
24. Any condition that makes the patient unable to complete the study within 3 months.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Glycemic Variability | 12 weeks
  Glycemic Variability defined by the mean amplitude of glycemic excursion (MAGE) measured by CGMS

SECONDARY OUTCOMES:
Glycated hemoglobin A1c (HbA1c) measured as percentage (%) | 12 weeks
  Glycated hemoglobin A1c (HbA1c) measured by HPLC (High Performance Liquid Chromatography)
Fasting plasma glucose (FPG) measured by hexokinase method (mg/dL) | 12 weeks
  Fasting plasma glucose (FPG) measured by hexokinase method after at least 8 hours in fasting state.
Postprandial glucose (PPG) measured by hexokinase method (mg/dL) | 12 weeks
  Postprandial glucose (PPG) measured by hexokinase method 2 hours after lunch
HbA1c ≤6.5% and <7% | 12 weeks
  Achievement of HbA1c ≤6.5% and <7% at the end of the study
Glycemic variability 2 | 12 weeks
  Glycemic variability defined by the interquartile range (IQR - interval between 25th and 75th percentiles) measured by CGMS
Glycemic variability 3 | 12 weeks
  Glycemic Variability defined by the Standard Deviation of the mean glycaemia (SD) measured by CGMS
Glycemic variability 4 | 12 weeks
  Glycemic Variability defined by the Coefficient of Variation (CV) measured by CGMS
Hypoglycemia | 12 weeks
  Time spent on hypoglycemic range (glycaemia <70mg/dL) measured by CGMS

CONTACTS AND LOCATIONS:
Overall Officials: Andre GD Vianna, MD, Principal Investigator — Centro de Diabetes Curitiba
Locations (1):
- Centro de Diabetes Curitiba, Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeFronzo RA, Hompesch M, Kasichayanula S, Liu X, Hong Y, Pfister M, Morrow LA, Leslie BR, Boulton DW, Ching A, LaCreta FP, Griffen SC. Characterization of renal glucose reabsorption in response to dapagliflozin in healthy subjects and subjects with type 2 diabetes. Diabetes Care. 2013 Oct;36(10):3169-76. doi: 10.2337/dc13-0387. Epub 2013 Jun 4. PMID 23735727
- [Background] Vasilakou D, Karagiannis T, Athanasiadou E, Mainou M, Liakos A, Bekiari E, Sarigianni M, Matthews DR, Tsapas A. Sodium-glucose cotransporter 2 inhibitors for type 2 diabetes: a systematic review and meta-analysis. Ann Intern Med. 2013 Aug 20;159(4):262-74. doi: 10.7326/0003-4819-159-4-201308200-00007. PMID 24026259
- [Background] Bailey CJ, Gross JL, Hennicken D, Iqbal N, Mansfield TA, List JF. Dapagliflozin add-on to metformin in type 2 diabetes inadequately controlled with metformin: a randomized, double-blind, placebo-controlled 102-week trial. BMC Med. 2013 Feb 20;11:43. doi: 10.1186/1741-7015-11-43. PMID 23425012
- [Background] Rosenstock J, Vico M, Wei L, Salsali A, List JF. Effects of dapagliflozin, an SGLT2 inhibitor, on HbA(1c), body weight, and hypoglycemia risk in patients with type 2 diabetes inadequately controlled on pioglitazone monotherapy. Diabetes Care. 2012 Jul;35(7):1473-8. doi: 10.2337/dc11-1693. Epub 2012 Mar 23. PMID 22446170
- [Background] Henry RR, Murray AV, Marmolejo MH, Hennicken D, Ptaszynska A, List JF. Dapagliflozin, metformin XR, or both: initial pharmacotherapy for type 2 diabetes, a randomised controlled trial. Int J Clin Pract. 2012 May;66(5):446-56. doi: 10.1111/j.1742-1241.2012.02911.x. Epub 2012 Mar 13. PMID 22413962
- [Background] ADVANCE Collaborative Group; Patel A, MacMahon S, Chalmers J, Neal B, Billot L, Woodward M, Marre M, Cooper M, Glasziou P, Grobbee D, Hamet P, Harrap S, Heller S, Liu L, Mancia G, Mogensen CE, Pan C, Poulter N, Rodgers A, Williams B, Bompoint S, de Galan BE, Joshi R, Travert F. Intensive blood glucose control and vascular outcomes in patients with type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2560-72. doi: 10.1056/NEJMoa0802987. Epub 2008 Jun 6. PMID 18539916
- [Background] Zhang CL, Katoh M, Shibasaki T, Minami K, Sunaga Y, Takahashi H, Yokoi N, Iwasaki M, Miki T, Seino S. The cAMP sensor Epac2 is a direct target of antidiabetic sulfonylurea drugs. Science. 2009 Jul 31;325(5940):607-10. doi: 10.1126/science.1172256. PMID 19644119
- [Background] Monnier L, Mas E, Ginet C, Michel F, Villon L, Cristol JP, Colette C. Activation of oxidative stress by acute glucose fluctuations compared with sustained chronic hyperglycemia in patients with type 2 diabetes. JAMA. 2006 Apr 12;295(14):1681-7. doi: 10.1001/jama.295.14.1681. PMID 16609090
- [Background] Kuenen JC, Borg R, Kuik DJ, Zheng H, Schoenfeld D, Diamant M, Nathan DM, Heine RJ; ADAG Study Group. Does glucose variability influence the relationship between mean plasma glucose and HbA1c levels in type 1 and type 2 diabetic patients? Diabetes Care. 2011 Aug;34(8):1843-7. doi: 10.2337/dc10-2217. Epub 2011 Jun 23. PMID 21700921
- [Background] Natali A, Ferrannini E. Endothelial dysfunction in type 2 diabetes. Diabetologia. 2012 Jun;55(6):1559-63. doi: 10.1007/s00125-011-2445-5. Epub 2012 Jan 20. PMID 22261897
- [Background] Bloomgarden ZT. Cardiovascular disease in diabetes. Diabetes Care. 2010 Apr;33(4):e49-54. doi: 10.2337/dc10-zb04. No abstract available. PMID 20351221
- [Background] Di Flaviani A, Picconi F, Di Stefano P, Giordani I, Malandrucco I, Maggio P, Palazzo P, Sgreccia F, Peraldo C, Farina F, Frajese G, Frontoni S. Impact of glycemic and blood pressure variability on surrogate measures of cardiovascular outcomes in type 2 diabetic patients. Diabetes Care. 2011 Jul;34(7):1605-9. doi: 10.2337/dc11-0034. Epub 2011 May 24. PMID 21610126
- [Background] Guerci B, Monnier L, Serusclat P, Petit C, Valensi P, Huet D, Raccah D, Colette C, Quere S, Dejager S. Continuous glucose profiles with vildagliptin versus sitagliptin in add-on to metformin: results from the randomized Optima study. Diabetes Metab. 2012 Oct;38(4):359-66. doi: 10.1016/j.diabet.2012.06.001. Epub 2012 Jul 17. PMID 22809630
- [Background] Marfella R, Barbieri M, Grella R, Rizzo MR, Nicoletti GF, Paolisso G. Effects of vildagliptin twice daily vs. sitagliptin once daily on 24-hour acute glucose fluctuations. J Diabetes Complications. 2010 Mar-Apr;24(2):79-83. doi: 10.1016/j.jdiacomp.2009.01.004. Epub 2009 Mar 4. PMID 19261490
- [Background] Service FJ, Molnar GD, Rosevear JW, Ackerman E, Gatewood LC, Taylor WF. Mean amplitude of glycemic excursions, a measure of diabetic instability. Diabetes. 1970 Sep;19(9):644-55. doi: 10.2337/diab.19.9.644. No abstract available. PMID 5469118
- [Background] Zaccardi F, Stefano PD, Busetto E, Federici MO, Manto A, Infusino F, Lanza GA, Pitocco D, Ghirlanda G. Group of signs: a new method to evaluate glycemic variability. J Diabetes Sci Technol. 2008 Nov;2(6):1061-5. doi: 10.1177/193229680800200614. PMID 19885294
- [Background] Bergenstal RM, Ahmann AJ, Bailey T, Beck RW, Bissen J, Buckingham B, Deeb L, Dolin RH, Garg SK, Goland R, Hirsch IB, Klonoff DC, Kruger DF, Matfin G, Mazze RS, Olson BA, Parkin C, Peters A, Powers MA, Rodriguez H, Southerland P, Strock ES, Tamborlane W, Wesley DM. Recommendations for standardizing glucose reporting and analysis to optimize clinical decision making in diabetes: the Ambulatory Glucose Profile (AGP). Diabetes Technol Ther. 2013 Mar;15(3):198-211. doi: 10.1089/dia.2013.0051. Epub 2013 Feb 28. PMID 23448694
- [Background] Inkster B, Zammitt NN, Frier BM. Drug-induced hypoglycaemia in type 2 diabetes. Expert Opin Drug Saf. 2012 Jul;11(4):597-614. doi: 10.1517/14740338.2012.694424. Epub 2012 Jun 13. PMID 22690846
- [Background] Nauck MA, Del Prato S, Meier JJ, Duran-Garcia S, Rohwedder K, Elze M, Parikh SJ. Dapagliflozin versus glipizide as add-on therapy in patients with type 2 diabetes who have inadequate glycemic control with metformin: a randomized, 52-week, double-blind, active-controlled noninferiority trial. Diabetes Care. 2011 Sep;34(9):2015-22. doi: 10.2337/dc11-0606. Epub 2011 Aug 4. PMID 21816980
- [Background] Jabbour SA, Hardy E, Sugg J, Parikh S; Study 10 Group. Dapagliflozin is effective as add-on therapy to sitagliptin with or without metformin: a 24-week, multicenter, randomized, double-blind, placebo-controlled study. Diabetes Care. 2014;37(3):740-50. doi: 10.2337/dc13-0467. Epub 2013 Oct 21. PMID 24144654
- [Background] Wilding JP, Woo V, Soler NG, Pahor A, Sugg J, Rohwedder K, Parikh S; Dapagliflozin 006 Study Group. Long-term efficacy of dapagliflozin in patients with type 2 diabetes mellitus receiving high doses of insulin: a randomized trial. Ann Intern Med. 2012 Mar 20;156(6):405-15. doi: 10.7326/0003-4819-156-6-201203200-00003. PMID 22431673
- [Background] Wilding JP, Woo V, Rohwedder K, Sugg J, Parikh S; Dapagliflozin 006 Study Group. Dapagliflozin in patients with type 2 diabetes receiving high doses of insulin: efficacy and safety over 2 years. Diabetes Obes Metab. 2014 Feb;16(2):124-36. doi: 10.1111/dom.12187. Epub 2013 Aug 29. PMID 23911013
- [Background] Plosker GL. Dapagliflozin: a review of its use in type 2 diabetes mellitus. Drugs. 2012 Dec 3;72(17):2289-312. doi: 10.2165/11209910-000000000-00000. PMID 23170914
- [Background] Drouin P, Standl E; Diamicron MR Study Group. Gliclazide modified release: results of a 2-year study in patients with type 2 diabetes. Diabetes Obes Metab. 2004 Nov;6(6):414-21. doi: 10.1111/j.1462-8902.2004.00404.x. PMID 15479217
- [Background] McGavin JK, Perry CM, Goa KL. Gliclazide modified release. Drugs. 2002;62(9):1357-64; discussion 1365-6. doi: 10.2165/00003495-200262090-00010. PMID 12076188
- [Background] Avogaro A. Treating diabetes today with gliclazide MR: a matter of numbers. Diabetes Obes Metab. 2012 Jan;14 Suppl 1:14-9. doi: 10.1111/j.1463-1326.2011.01508.x. PMID 22118706
- [Background] Lin SD, Wang JS, Hsu SR, Sheu WH, Tu ST, Lee IT, Su SL, Lin SY, Wang SY, Hsieh MC. The beneficial effect of alpha-glucosidase inhibitor on glucose variability compared with sulfonylurea in Taiwanese type 2 diabetic patients inadequately controlled with metformin: preliminary data. J Diabetes Complications. 2011 Sep-Oct;25(5):332-8. doi: 10.1016/j.jdiacomp.2011.06.004. Epub 2011 Aug 2. PMID 21813293
- [Background] Czerwoniuk D, Fendler W, Walenciak L, Mlynarski W. GlyCulator: a glycemic variability calculation tool for continuous glucose monitoring data. J Diabetes Sci Technol. 2011 Mar 1;5(2):447-51. doi: 10.1177/193229681100500236. PMID 21527118
- [Background] Hill NR, Oliver NS, Choudhary P, Levy JC, Hindmarsh P, Matthews DR. Normal reference range for mean tissue glucose and glycemic variability derived from continuous glucose monitoring for subjects without diabetes in different ethnic groups. Diabetes Technol Ther. 2011 Sep;13(9):921-8. doi: 10.1089/dia.2010.0247. Epub 2011 Jun 29. PMID 21714681